CLINICAL TRIAL: NCT07223515
Title: Effectiveness of Four Amniotic Membrane-based Skin Substitute Allografts Added to Standard Care in Chronic Diabetic Foot Ulcers, Venous Leg Ulcers, and Pressure Ulcers (HEAL-4): A Multi-Site Real-World Study
Brief Title: HEAL-4: Real-World Effectiveness of 4 Amniotic Allografts Adjunctive to Standard Care in DFU, VLU, and PU
Acronym: HEAL-4
Status: Active, not recruiting | Type: Observational
Sponsor: Dynamic Medical Services dba Acesso Biologics (Industry)
Responsible Party: Sponsor
Other Study IDs: AB-RWE-2025-01
Record Dates: First submitted 2025-09-19; First posted 2025-11-03 (Actual); Last update posted 2025-11-03 (Actual); Status verified 2025-10

CONDITIONS: Diabetic Foot Ulcer (DFU); Venous Leg Ulcers (VLUs); Pressure Ulcers, Bedsores, Decubitus Ulcer
MeSH Terms: conditions — Diabetic Foot; Pressure Ulcer

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective

GROUPS / COHORTS (15):
- Acesso DL + Standard care for DFU: Patients who received Acesso DL plus standard care for their DFU
- Acesso TL + Standard care for DFU: Patients who received Acesso TL plus standard care for their DFU
- Neostim DL + Standard care for DFU: Patients who received Neostim DL plus standard care for their DFU
- Neostim TL + Standard care for DFU: Patients who received Neostim TL plus standard care for their DFU
- Standard care alone for DFU: Patients who received standard care only for their DFU
- Acesso DL + Standard care for VLU: Patients who received Acesso DL plus standard care for their VLU
- Acesso TL + Standard care for VLU: Patients who received Acesso TL plus standard care for their VLU
- Neostim DL + Standard care for VLU: Patients who received Neostim DL plus standard care for their VLU
- Neostim TL + Standard care for VLU: Patients who received Neostim TL plus standard care for their VLU
- Standard care alone for VLU: Patients who received standard care only for their VLU
- Acesso DL + Standard care for PU: Patients who received Acesso DL plus standard care for their PU
- Acesso TL + Standard care for PU: Patients who received Acesso TL plus standard care for their PU
- Neostim DL + Standard care for PU: Patients who received Neostim DL plus standard care for their PU
- Neostim TL + Standard care for PU: Patients who received Neostim TL plus standard care for their PU
- Standard care alone for PU: Patients who received standard care only for their PU

SUMMARY:
This retrospective multi-site observational cohort study uses electronic health records (EHR) from U.S. wound care centers to evaluate the effectiveness of four amniotic membrane allografts (Acesso DL, Acesso TL, Neostim DL, Neostim TL) when added to standard wound care for diabetic foot ulcers (DFU), venous leg ulcers (VLU), and pressure ulcers (PU). The primary endpoint is complete wound closure by 12 weeks. Secondary outcomes include time-to-closure, ≥50% wound-area reduction at 4 weeks, wound-related complications (infection, hospitalization, emergency department visits, and major/minor amputation).

ELIGIBILITY:
Inclusion Criteria:

* Adults ≥18; DFU/VLU/PU; sufficient observability

Exclusion Criteria:

* Non-study advanced biologic product use within 60 days pre-index; insufficient follow-up

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with DFU, VLU, or PU
Sampling Method: Non-Probability Sample
Enrollment: 2000 (Estimated)
Dates: Start 2025-10-24 (Actual); Primary Completion 2025-11 (Estimated); Study Completion 2025-11 (Estimated)

PRIMARY OUTCOMES:
Complete wound closure at 12 Weeks | From index visit to 12 weeks post-index
  Proportion of index wounds with 100% epithelialization, no drainage or dressings; confirmation on ≥1 follow-up within 60 days

SECONDARY OUTCOMES:
Time to complete wound closure | From index visit up to 24 months post-index
  Time from the index visit to primary complete wound closure for wounds that heal during the study period
≥50% wound area reduction at 4 weeks | From index visit to 4 weeks post-index
  Proportion of patients whose wounds close greater than 50% within 4 weeks from the index visit
Wound-related complications | From index visit up to 24 months post-index
  Wound-related complications including infection requiring treatment, hospitalization, ED visits, and major or minor amputation

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Optalis, Novi, Michigan
  - ProCure Health, Murfreesboro, Tennessee